CLINICAL TRIAL: NCT02948634
Title: A Prospective, Randomized, Double-blind, Sham-controlled Study of the Low-level Phoenix Thera-lase 42 Watt Laser in Patients With Chronic Fibromyalgia
Brief Title: Low-level Laser Therapy in Patients With Chronic Fibromyalgia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU 072016-079
Record Dates: First submitted 2016-10-19; First posted 2016-10-28 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Phoenix Laser Treatment (Sham Comparator): Each participant will receive a series of nine active laser or sham treatments on a M-W-F schedule over the three week treatment period. Sham treatment will be delivered via the same protocol in terms of time, application, and areas of treatment as stated above, except the laser unit will not discharge any photonic energy.
  Interventions: Device: Sham Phoenix Laser Treatment
- Active Phoenix Laser Treatment (Active Comparator): Each participant will receive a series of nine active laser or sham treatments on a M-W-F schedule over the three week treatment period. Participants in the laser treatment group will be treated at 42 watts for up to 60 seconds at tender spots in the spine or extremities. Total treatment time is not to exceed 30 minutes.
  Interventions: Device: Active Phoenix Laser Treatment

INTERVENTIONS:
Device: Sham Phoenix Laser Treatment — Sham treatment will be delivered via the same protocol in terms of time, application, and areas of treatment as stated above, except the laser unit will not discharge any photonic energy. Intervention will take place in the therapy room at the McDermott Center for Pain Management, which is appropriately equipped for laser administration. Application of therapeutic laser will be completed by licensed physical therapists who have completed safety training for therapeutic laser application including appropriate use of safety eyewear, room access, laser signage for laser use, and patient monitoring.
  Arms: Sham Phoenix Laser Treatment
Device: Active Phoenix Laser Treatment — The 30 min treatments will include multiple 60 sec applications to all tender points on the spine or extremities and a 10 minute application along the bilateral sympathetic ganglion in the paraspinous region. The treatment will be applied via a non-contact method, with the laser applicator held 12-18 inches above the participant's skin.
  Arms: Active Phoenix Laser Treatment

SUMMARY:
The purpose of this study is to examine the use of low level therapeutic laser (LLLT) for its effects on pain, fatigue, and physical function in individuals with fibromyalgia.

DETAILED DESCRIPTION:
Fifty consenting participants with long-standing fibromyalgia (> 3 mo duration) will be randomized to one of two treatment groups (n=25 per group) according to a computer generated randomization table. Group 1 will be the 'sham' control group and Group 2 will be the 'active' laser treatment group. The study will be conducted in a double-blind fashion using a standard 42 watt Class IV laser which has a switch at the back of the device which allows the laser to operate in the 'inactive' mode despite giving the operator and patients the appearance of being active (e.g., generates skin warmth and a red beam of light). Treatment will be administered three times/week for three weeks. Data will be collected across the 3-week intervention and one week after completion of the intervention. Data will be analyzed with appropriate statistical methods.

The following outcome measures will be collected at baseline: (1)Standardized SF-36 questionnaire; (2) Symptom Impact Questionnaire; (3) current analgesic medication usage; (4) pressure-pain threshold testing over tender points; and (5) spinal range of motion with an inclinometer and accelerometer. Outcome measures (2) and (3) will be re-assessed during the treatment phase at the end of weeks 1, 2 and 3. At 1 week and 1 month after the last laser/sham treatment session, all baseline assessments will be repeated, in addition to a global rating of change scale. Any patient who reports any harm from the laser/sham treatments on the helpfulness scale will be queried for specific harm details.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old
2. Pre-existing medical conditions are under stable control
3. Diagnosis of fibromyalgia by Widespread Pain Index and Symptom Severity Score
4. Able to wear laser protective eyewear during the treatment session
5. Ability to speak English and complete testing

Exclusion Criteria:

1. Presence of another pain syndrome that has anatomical overlapping with fibromyalgia pain
2. Unstable psychiatric disorders or cognitive dysfunction or serious memory impairment
3. Previous treatment with low level laser therapy
4. Contraindication to receiving laser treatments
5. Current use of photosensitive medication (has been instructed to minimize sun exposure)
6. Active metastasis
7. Active infection
8. Impaired sensation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Zafereo, PT, PhD, Principal Investigator — UT Southwestern
Locations (1):
- McDermott Pain Management Clinic, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham Phoenix Laser Treatment | Active Phoenix Laser Treatment
Started | 17 | 11
Completed | 7 | 9
Not Completed | 10 | 2
Not completed — Lack of efficacy and study suspended | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Phoenix Laser Treatment | Active Phoenix Laser Treatment | Total
Number analyzed (Participants) | 17 | 11 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (10.3) | 53.0 (10.2) | 53.0 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: percent]
  % white | 75 | 75 | 75
  % black | 25 | 25 | 25
Revised Symptom Impact Questionnaire [Mean (Standard Deviation); unit: units on a scale] | 62.0 (7.6) | 68.3 (14.8) | 65.7 (12.5)

OUTCOME MEASURES:

1. Primary Outcome: The Revised Symptom Impact Questionnaire
Description: Self-Report Questionnaire containing 21 questions, maximum/worse score=100; minimum/best score=0.
Time Frame: baseline, 1 week, and 1 month after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Phoenix Laser Treatment | Active Phoenix Laser Treatment
Number analyzed (Participants) | 7 | 9
score on a scale
  Baseline | 62.0 (7.6) | 68.3 (14.8)
  1 week | 47.1 (21.8) | 50.5 (22.5)
  1 month | 45.8 (22.5) | 50.2 (25.3)
Statistical Analysis 1: Comparison: Sham Phoenix Laser Treatment vs Active Phoenix Laser Treatment; Test type: Superiority; p = 0.43, ANOVA

2. Secondary Outcome: RAND 36-Item Health Survey
Description: Pain Domain: 2 Questions, 0 minimum/worse score, 100 maximum/best score
Time Frame: baseline, 1 week, and 1 month after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Phoenix Laser Treatment | Active Phoenix Laser Treatment
Number analyzed (Participants) | 7 | 9
score on a scale
  Baseline | 27.2 (13.0) | 27.2 (15.2)
  1 week | 33.6 (2.7) | 37.8 (20.6)
  1 month | 41.8 (5.5) | 36.4 (22.6)
Statistical Analysis 1: Comparison: Sham Phoenix Laser Treatment vs Active Phoenix Laser Treatment; Test type: Superiority; p = 0.32, ANOVA

3. Secondary Outcome: Global Rating of Change Scale
Description: Self report tool describing the degree of change since baseline. Minimum/worse value is -7. Maximum/best value is +7.
Time Frame: 1 week and 1 month after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Phoenix Laser Treatment | Active Phoenix Laser Treatment
Number analyzed (Participants) | 7 | 9
score on a scale
  1 week | 0.4 (3.3) | 2.8 (2.0)
  1 month | 0 (3.1) | 1.3 (3.9)
Statistical Analysis 1: Comparison: Sham Phoenix Laser Treatment vs Active Phoenix Laser Treatment; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Sham Phoenix Laser Treatment | Active Phoenix Laser Treatment
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/11
Other Adverse Events (participants affected / at risk) | 0/17 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT02948634/Prot_SAP_000.pdf